CLINICAL TRIAL: NCT01110564
Title: A Cross-sectional Observational Study to Investigate Daily Symptom Variability, Effects of Symptom on Morning Activities and Therapeutic Expectations of Patients and Physicians in Chronic Obstructive Pulmonary Disease - SUNRISE Study
Brief Title: Study to Investigate Daily Symptom Variability, Symptom Effects on Morning Activities of Chronic Obstructive Disease
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstrraZeneca
Other Study IDs: NIS-RTR-DUM-2009/1
Record Dates: First submitted 2010-04-23; First posted 2010-04-26 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; daily symptom variability; effects of symptom on morning activities
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- 1: COPD patients

SUMMARY:
The primary objective of this non-interventional study is to evaluate daily symptom variability in COPD patients. The secondary objectives are; to evaluate effects of COPD symptoms on the morning activities of patients, to determine therapeutic expectations of patients and physicians in COPD, to determine which and how frequent non-drug approaches are recommended in order to prevent COPD exacerbations, to define COPD patient profiles about the below-mentioned issues: Demographic characteristics, Disease characteristics, Concomitant diseases and implemented drug treatments. All patients, who apply to the study physicians and fulfill all patient selection criteria during patient enrolment period, will be included. Patients, who provide all of the following measures will be included in the study: To apply to a physician for outpatient treatment for any reason, Age over 45 years, being diagnosed with COPD, being a smoker or used to be a smoker once (> 10 package years), to give consent for the use of their medical data. The patients that exhibit the following exclusion criteria will be excluded from the study: COPD exacerbations still on-going or experienced in the last 3 months (Exacerbation is defined as worsening of COPD symptoms leading to antibiotic and/or short-term oral steroid treatment and/or hospitalization or admission to the emergency unit.); Presence of lung cancer or an important respiratory disease such as bronchiectasis, pulmonary fibrosis, interstitial pulmonary disease, tuberculosis, sarcoidosis; Participation in an interventional clinical trial at present and Enrollment in this study once. In this study, patients will be recorded at their visit to the physician and there will be no follow-up thereafter.

ELIGIBILITY:
Inclusion Criteria:

* To apply to a physician for outpatient treatment for any reason; being diagnosed with COPD
* being a smoker or used to be a smoker once (> 10 package years)
* to give consent for the use of their medical data

Exclusion Criteria:

* COPD exacerbations still on-going or experienced in the last 3 months
* Presence of lung cancer or an important respiratory disease such as bronchiectasis, pulmonary fibrosis, interstitial pulmonary disease, tuberculosis, sarcoidosis
* Participation in an interventional clinical trial at present and Enrollment in this study once

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Obstructive Pulmonary Disease (COPD)
Sampling Method: Non-Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To evaluate daily symptom variability in Chronic Obstructive Pulmonary Disease (COPD) patients | April - Dec 2010

SECONDARY OUTCOMES:
To evaluate effects of COPD symptoms on the morning activities of patients; To determine therapeutic expectations of patients and physicians in COPD | April - Dec 2010
To define COPD patient profiles about the below-mentioned issues: Demographic characteristics; Disease characteristics; Concomitant diseases; Implemented drug treatments | April - Dec 2010
To determine which and how frequent non-drug approaches are recommended in order to prevent COPD exacerbations | April - Dec 2010

CONTACTS AND LOCATIONS:
Overall Officials: Tulin Kuyucu, Study Chair — Sureyyapasa Chest Disease Hospital
Locations (19):
- Turkey (Türkiye) (19):
  - Research Site, Aksaray
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Aydin
  - Research Site, Bilecik
  - Research Site, Bolu
  - Research Site, Bursa
  - Research Site, Denizli
  - Research Site, Elâzığ
  - Research Site, Hatay
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kocaeli
  - Research Site, Konya
  - Research Site, Manisa
  - Research Site, Rize
  - Research Site, Samsun
  - Research Site, Sanliurfa
  - Research Site, Yozgat